CLINICAL TRIAL: NCT06045013
Title: Comparison of the Efficacy Between Ultrasound-guided Dextrose Injection Versus Dextrose With Methylprednisolone Injection in Patients With Carpal Tunnel Syndrome: a Prospective, Randomized Double-blind Clinical Trial.
Brief Title: Ultrasound-guided Dextrose Injection Versus Dextrose With Methylprednisolone in Carpal Tunnel Syndrome
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: General and Veteran Hospital Croatian Pride Knin (Other)
Collaborators: Clinical Hospital Centre Zagreb (Other); School of Public Health Andrija Štampar (Unknown)
Responsible Party: Principal Investigator, Igor Begović, Physical medicine and rehabilitation specialist, General and Veteran Hospital Croatian Pride Knin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 510.01/23-01/76
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; Ultrasonography; Injections; Glucose; Glucocorticoids; Pain; Functional Status; Hand Strength, Quality of Life
MeSH Terms: conditions — Carpal Tunnel Syndrome; Pain | interventions — Glucose; Methylprednisolone Acetate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 5% dextrose injection (Active Comparator): Ultrasound-guided 4 ml single injection of 5% dextrose
  Interventions: Drug: 5% dextrose injection
- 5% dextrose injections with methylprednisolone acetate (Active Comparator): Ultrasound-guided single injection of 3 ml 5% dextrose plus 1 ml 40 mg/ml methylprednisolone acetate
  Interventions: Drug: 5% dextrose injections with methylprednisolone acetate 40 mg/ml

INTERVENTIONS:
Drug: 5% dextrose injection — Single ultrasound-guided injection of 4 ml 5% dextrose in carpal tunnel via ulnar approach.
  Other Names: 5% dextrose
  Arms: 5% dextrose injection
Drug: 5% dextrose injections with methylprednisolone acetate 40 mg/ml — Single ultrasound-guided injection of 3 ml 5% dextrose with 1 ml 40 mg/ml methylprednisolone acetate in carpal tunnel via ulnar approach.
  Other Names: Depo-Medrol 40 mg/ml
  Arms: 5% dextrose injections with methylprednisolone acetate

SUMMARY:
The goal of this prospective, randomized, double-blinded, head-to-head comparative study is to compare the efficacy of ultrasound-guided 4 ml 5% dextrose perineural injection versus 3 ml 5% dextrose with 1 ml 40 mg/ml methylprednisolone perineural injection in patients with carpal tunnel syndrome (CTS).

The main questions it aims to answer are:

Is there a difference in efficacy between interventions regarding 1. pain alleviation, 2. improvement in symptoms severity and functional status, 3. improvement in grip strength, 4. size of median nerve cross-sectional area, and 5. improvement in quality of life during the six-month post-intervention follow-up period?

DETAILED DESCRIPTION:
The research will be conducted in the General and Veteran Hospital "Croatian Pride" Knin.

The research will be a prospective, randomized, double-blinded, head-to-head comparative study.

The goal of the research is to compare the efficacy of ultrasound-guided 5% dextrose injection versus 5% dextrose with 40 mg methylprednisolone injection in patients with carpal tunnel syndrome (CTS).

Randomization of patients will be performed before the intervention using computer software.

All participants will sign written informed consent and the study will be performed under the ethical standards as laid down in the 1964 Declaration of Helsinki and its later amendments or comparable ethical standards. The study is approved by the Ethical Committee at the General and Veteran Hospital "Croatian Pride" Knin (approval number: 510.01/23-01/79).

Adult participants aged between 18 and 80 years with a clinical and electrophysiological diagnosis of idiopathic CTS referred to the Physical Medicine and Rehabilitation clinic will be randomly assigned into two groups using a random number generating software in a 1:1 manner.

Since patients can have CTS in one or both hands, randomization will be conducted according to the patient, thus the same patient can receive the intervention only on one side which will be considered worst.

The minimum sample size of a total of 70 participants (35 in each group) was estimated by analyzing the power of the t-test for independent samples according to the following characteristics: type one error (α=0.05), power (1-ß=0.80), and effect size (d=0.68).

The power analysis of the test was performed using the computer program G*Power for Windows, version 3.1.3.

IBM SPSS Statistics version 29.0 software will be used for the data analysis.

Group one will receive an ultrasound-guided 4 ml single perineural injection of 5% dextrose in the carpal tunnel and group two ultrasound-guided single perineural injection of 3 ml 5% dextrose plus 1 ml 40 mg/ml methylprednisolone acetate in the carpal tunnel.

Participants, the physician who will perform the injection procedure and the assessor will be blinded for the treatment allocation. The only person who will know which intervention drug it is about will be the nurse who will prepare the medicine according to the randomization.

Clinical diagnosis of CTS will be made in the presence of at least one symptom (1. pain, 2. pricking, 3. tingling, 4. burning, or 5. numbness in the innervation area of the median nerve on the hand) and at least one sign (1. objective disturbance of the sense of touch, i.e. hypoesthesia or dysesthesia in the innervation area of the median nerve on the hand, 2. positive Tinel's sign, 3. positive Phalen's sign, or 4. positive compression test).

Inclusion criteria are age between 18 and 80 years and the diagnosis of idiopathic CTS based on clinical and electrophysiological criteria.

Exclusion criteria are contraindications for local application of methylprednisolone or 5% dextrose (hypersensitivity to the drug, infection, and skin damage at the application site), previous wrist surgery, traumatic wrist injury within 2 years, previous wrist injection within 6 months, previous physical therapy within 6 months, history of traumatic peripheral nerve injury in the upper extremity, brachial plexopathy, severe cervical radiculopathy and thoracic outlet syndrome, history of diabetes, history of thyroid disease, history of inflammatory rheumatic disease, pregnancy and inability to cooperate with the study protocol.

Basic demographic data will be obtained: gender, age, Body Mass Index (BMI), level of education, occupation, rating of hand activity and force level applied on the hand during the day, cigarette smoking, hand dominance, affected hand, symptom duration, and history of comorbid conditions.

Pain intensity (using a 10 cm Visual Analogue Scale; VAS pain, 0-10; 0=no pain, 10=the most severe pain), symptoms severity and functional impairment (using the Boston Carpal Tunnel Questionnaire; BCTQ), grip strength (using the Jamar hydraulic hand dynamometer in kilograms), median nerve cross-sectional area (CSA) (using diagnostic ultrasound at the carpal tunnel inlet), and quality of life (QoL) (using 36-Item Short Form Survey; SF-36) will be measured immediately before injection, at 4, 12, and 24 weeks post-injection.

The primary outcome measure will be the change in pain intensity at 4 weeks post-injection.

Secondary outcome measures will be the change in pain intensity at 12 and 24 weeks post-injection, and the changes in symptoms severity and functional impairment, grip strength, median nerve CSA, and QoL at 4, 12, and 24 weeks post-injection.

During the study, acetaminophen and tramadol will be allowed for occasional pain relief except for two days prior to the evaluation sessions due to possible interference with the results.

Physical therapy, use of wrist splints, acupuncture, and invasive interventions for CTS other than those included in the study protocol will not be allowed during the study.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years,
* the diagnosis of idiopathic CTS.

Exclusion Criteria:

* contraindications for local application of methylprednisolone or 5% dextrose (hypersensitivity to the drug, infection and skin damage at the application site),
* previous wrist surgery,
* traumatic wrist injury within 2 years,
* previous wrist injection within 6 months,
* previous physical therapy within 6 months,
* history of peripheral traumatic nerve injury in the upper extremity, brachial plexopathy, severe cervical radiculopathy, and thoracic outlet syndrome,
* history of diabetes
* history of thyroid disease,
* history of inflammatory rheumatic disease,
* pregnancy,
* inability to cooperate with the study protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity at 4 weeks post injection | before injection, 4 weeks post injection
  Assessment of pain intensity using 10 cm Visual Analogue Scale (VAS pain), 0-10; 0=no pain, 10=the most severe pain.

SECONDARY OUTCOMES:
Pain intensity at 12 and 24 weeks post injection | before injection,12 and 24 weeks post injection.
  Assessment of pain intensity using 10 cm Visual Analogue Scale (VAS pain), 0-10; 0=no pain, 10=the most severe pain.
Symptoms severity and functional impairment of carpal tunnel syndrome (CTS) | before injection, 4, 12 and 24 weeks post injection.
  Assessment of CTS symptoms severity and functional impairment using the Boston Carpal Tunnel Questionnaire (BCTQ).
Grip strength | before injection, 4, 12 and 24 weeks post injection.
  Assessment of grip strength using the Jamar hydraulic hand dynamometer in kilograms.
Median nerve cross-sectional area (CSA) | before injection, 4, 12 and 24 weeks post injection.
  The CSA of the median nerve measured by diagnostic ultrasound at the level of carpal tunnel.
Quality of life (QoL) | before injection, 4, 12 and 24 weeks post injection.
  Assessment of QoL using 36-Item Short Form Survey (SF-36).

CONTACTS AND LOCATIONS:
Overall Officials: Igor Begović, MD, Principal Investigator — General and Veteran Hospital "Croatian Pride" Knin, Croatia
Locations (1):
- General and Veteran Hospital "Croatian Pride" Knin, Knin, Croatia

REFERENCES:
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823
- [Background] Gao N, Yan L, Ai F, Kang J, Wang L, Weng Y. Comparison of the Short-Term Clinical Effectiveness of 5% Dextrose Water, Platelet-rich Plasma and Corticosteroid Injections for Carpal Tunnel Syndrome: A Systematic Review and Network Meta-analysis of Randomized Controlled Trials. Arch Phys Med Rehabil. 2023 May;104(5):799-811. doi: 10.1016/j.apmr.2022.11.009. Epub 2022 Dec 16. PMID 36529261
- [Background] Lin MT, Liao CL, Hsiao MY, Hsueh HW, Chao CC, Wu CH. Volume Matters in Ultrasound-Guided Perineural Dextrose Injection for Carpal Tunnel Syndrome: A Randomized, Double-Blinded, Three-Arm Trial. Front Pharmacol. 2020 Dec 17;11:625830. doi: 10.3389/fphar.2020.625830. eCollection 2020. PMID 33391002
- [Background] Levine DW, Simmons BP, Koris MJ, Daltroy LH, Hohl GG, Fossel AH, Katz JN. A self-administered questionnaire for the assessment of severity of symptoms and functional status in carpal tunnel syndrome. J Bone Joint Surg Am. 1993 Nov;75(11):1585-92. doi: 10.2106/00004623-199311000-00002. PMID 8245050
- [Background] Klauser AS, Halpern EJ, De Zordo T, Feuchtner GM, Arora R, Gruber J, Martinoli C, Loscher WN. Carpal tunnel syndrome assessment with US: value of additional cross-sectional area measurements of the median nerve in patients versus healthy volunteers. Radiology. 2009 Jan;250(1):171-7. doi: 10.1148/radiol.2501080397. Epub 2008 Nov 26. PMID 19037017
- [Background] Elnady B, Rageh EM, Ekhouly T, Fathy SM, Alshaar M, Fouda ES, Attar M, Abdelaal AM, El Tantawi A, Algethami MM, Bong D. Diagnostic potential of ultrasound in carpal tunnel syndrome with different etiologies: correlation of sonographic median nerve measures with electrodiagnostic severity. BMC Musculoskelet Disord. 2019 Dec 29;20(1):634. doi: 10.1186/s12891-019-3010-5. PMID 31884951
- See also: Randomization of patients into two groups will be carried out with the help of the above-listed web application. — https://www.randomizer.org/